CLINICAL TRIAL: NCT05697497
Title: A Brief Digital Exercise Program to Improve Physical Function Among Older Adults
Brief Title: Functional Activity Strength Training
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Professor and Vice Chair for Research Affairs, Department of Medicine, Penn State Health Milton S Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00016054
Record Dates: First submitted 2022-02-08; First posted 2023-01-26 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Walking, Difficulty
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: A delayed treatment control group will be used to compare the effects of the intervention to a control group. Both groups will complete their study visits at baseline, week 6, and week 12, with the intervention group starting their exercises immediately after the baseline visit and the delayed treatment control group starting their exercise intervention after their week 12 visit.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Condition (Experimental): The exercise intervention consists of a 4 minute daily routine that includes 2 upper body and 2 lower body exercises.
  Interventions: Behavioral: Daily exercise intervention
- Delayed-Treatment Control Group (No Intervention): The exercise intervention consists of a 4 minute daily routine that includes 2 upper body and 2 lower body exercises. Participants in the this arm will not start the exercise intervention until the day after the week 12 assessment.

INTERVENTIONS:
Behavioral: Daily exercise intervention — Participants will complete four exercises each day, The first two weeks they will be instructed to complete as many repetitions as possible, each day, for 15 seconds and progressing to 30 seconds per exercise after the first two weeks. Participants are asked to increase their goal repetitions by 1 or 2 from their previous best each week. For all exercises with modifications, we will encourage participants to move to the next most difficult modification once they can do 15 repetitions of that exercise.
  Arms: Intervention Condition

SUMMARY:
This study is a randomized trial of 100 older adults with mobility disability, who performed a similar brief daily, resistance training program. The investigators set out to answer the following question "Will a digital, brief daily exercise program be feasible, acceptable, and effective among older adults with walking limitations?" To answer that question, participants were assigned to an intervention or delayed-treatment control group. Intervention participants were assigned to complete two 30-second lower body exercises and two 30-second upper body exercises. Fitness tests were completed remotely three times during the 12-weeks (i.e., at baseline, week 6, week 12).

DETAILED DESCRIPTION:
This is a 12-week delayed-control randomized trial to answer the following question "Will a digital, brief daily exercise program be feasible, acceptable, and effective among older adults with walking limitations?" Participants who screen eligible will be assigned to one of four conditions, an immediate workout group, an immediate workout group with activity monitor, a delayed workout group or a delayed workout group with activity monitor. Participants will complete a daily 4-minute exercise routine at home and to record their results using an electronic survey. Other outcome measurements will be conducted remotely at baseline, 6, and 12 weeks.

The investigators hypothesize that participants in the AMRAP condition will report significant reductions in functional physical limitations, increased gait speed, and increased physical performance (i.e., increased exercise repetitions) from baseline to 6 weeks compared to those randomized to the delayed-treatment control.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* Difficulty with walking
* Providers must provide consent for their patient
* Access to the internet
* Must have a camera on computer, tablet, or smartphone
* Fluent in Egnlish

Exclusion Criteria:

* Chest pain or a heart condition on the PAR-Q
* Planning to have surgery in the next 3 months
* Cognitive impairment
* Unable to exercise
* Being currently physically active

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
30-Second Chair Stand | Baseline
  Leg strength and endurance test - number of chair stand repetitions in 30 seconds
30-Second Chair Stand | 6 weeks
  Leg strength and endurance test - number of chair stand repetitions in 30 seconds
30-Second Chair Stand | 12 weeks
  Leg strength and endurance test - number of chair stand repetitions in 30 seconds
Five Time Sit to Stand Test (5TSTS) | Baseline
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements. The score is the amount of time (to the nearest decimal in seconds) it takes a patient to transfer from a seated to a standing position and back to sitting five times.
Five Time Sit to Stand Test (5TSTS) | 6 weeks
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements. The score is the amount of time (to the nearest decimal in seconds) it takes a patient to transfer from a seated to a standing position and back to sitting five times.
Five Time Sit to Stand Test (5TSTS) | 12 weeks
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements. The score is the amount of time (to the nearest decimal in seconds) it takes a patient to transfer from a seated to a standing position and back to sitting five times.
Single Leg Stance Test (SLS) | 12 weeks
  Assessment of static postural and balance control.
Functional limitations | 12 weeks
  Physical Functioning Questionnaire from the National Health and Nutrition Examination Survey
Falls | 12 weeks
  Falls over the past 3 months will be assessed using the Behavioral Risk Factor Surveillance System survey.

SECONDARY OUTCOMES:
Walking gait cadence | 10 day period pre and post intervention
  Gait cadence will be measured in 50% of the participants using an activPAL device.
Pain on the Patient Reported Outcomes Measurement Information System (PROMIS) survey | 12 weeks
  Survey using questions from the NIH-supported Patient Reported Outcomes Measurement Information System (PROMIS). The minimal value for pain interference is not at all, while the minimum value for pain intensity is no pain. The maximum value for pain interference is very much, while the maximum value for pain intensity is worst pain imaginable. A higher score generally means a worse outcome.
Fatigue on the Patient Reported Outcomes Measurement Information System (PROMIS) survey | 12 weeks
  Survey using questions from the NIH-supported Patient Reported Outcomes Measurement Information System (PROMIS). The minimum value for fatigue is not at all, while the maximum value is very much. A higher score generally means a worse outcome.
Self-Efficay for Physical Activity (SEPA) | 12 weeks
  5-item measure that assesses an individual's confidence for engaging in exercise in the presence of barriers.
Percent of sessions attended | 12 weeks
  Patients will be considered adherent to the intervention when they enter their daily exercise performance data via daily survey. The percent of sessions attended will be calculated by dividing the number of sessions attended by the total number of sessions offered and multiplying the result by 100.
Heart rate | 12 weeks
  resting and maximal heart rates will be collected during the maximal exercise performance tests

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States